CLINICAL TRIAL: NCT06099717
Title: Clinical Performance of a Novel Implant-supported Fixed Dental Prostheses (iFDP): the Dual-cantilevered Single-implant Bridge (T-bridge)
Brief Title: Clinical Performance of Dual-cantilevered Single-implant Bridge
Acronym: T-bridge
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Collaborators: ITI International Team for Implantology, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Dual-cantilever single-implant
Record Dates: First submitted 2023-10-19; First posted 2023-10-25 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Dental Implant Failed
Keywords: Dental implant

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Who Masked: Investigator
Masking Description: Group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test (Experimental): Dual-cantilevered single implant bridge
  Interventions: Device: Dual-cantilevered implant bridge
- Control (Active Comparator): 3-unit implant fixed dental prosthesis
  Interventions: Device: 3-unit iFDP

INTERVENTIONS:
Device: Dual-cantilevered implant bridge — A 3-unit supported by one implant in the middle
  Arms: Test
Device: 3-unit iFDP — 3-unit fixed dental prosthesis supported by two implants
  Arms: Control

SUMMARY:
The study aims to evaluate the clinical performance (implant and prosthetic survival/ success rates) of a novel implant-supported fixed dental prosthesis design: the dual-cantilevered single implant bridge (T-Bridge) made out of monolithic zirconia bonded to a titanium base abutment (Variobase abutments)

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 20 years
* Willingness to sign an informed consent and participate in the study
* Three missing adjacent teeth in the posterior site.
* Tooth gap of 21-24 mm.
* Presence of natural or artificial opposing dentition
* Sufficient vertical interocclusal space of an implant restoration (7mm)
* Sufficient ridge height to place an implant of 10mm in length
* Sufficient ridge width for the placement of a 4.1mm diameter implant. Simultaneous GBR to achieve a width of 6.5mm will be included.

Exclusion Criteria:

* Any physical or mental disorder that would interfere with the ability to perform adequate oral hygiene or the capability of providing written informed consent and compliance with the protocol
* Any disorder that would interfere with wound healing or represent a contraindication for implant surgery, such as but not limited to uncontrolled diabetes or conditions resulting in or requiring immunosuppression, radiation, chemotherapy, frequent use of antibiotics or antiresorptive medication such as bisphosphonates.
* Pregnancy or lactation
* Heavy smoking habit with ≥ 10 cig/d
* Severe bruxism or clenching habits, presence of oro-facial pain
* Insufficient ridge width/height for the study implant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-06-30 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Implant and prosthetic success | 10 years
  Primary outcome parameter: implant and prosthetic success
  Implant success and survival rate will be defined according to established criteria (Buser et al. 1991):
  A surviving implant and/or restoration is defined as are in place at the time of the follow-up.
Implant and prosthetic survival | 10 years
  Implant success and survival rate will be defined according to established criteria (Buser et al. 1991): A surviving implant and/or restoration is defined as are in place at the time of the follow-up.

SECONDARY OUTCOMES:
Implant and prosthetic complications | 10 years
  Biological and/or Technical Implant and prosthetic complications

CONTACTS AND LOCATIONS:
Overall Officials: Martin Schimmel, Prof, Study Chair — University of Bern
Locations (1):
- Universidade Federal de Goias, Goiânia, Goiás, Brazil

IPD SHARING:
Plan to Share IPD: No